CLINICAL TRIAL: NCT02602457
Title: Exercise Training in Patients With Atrial Fibrillation (OPPORTUNITY Study)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20150427
Record Dates: First submitted 2015-11-03; First posted 2015-11-11 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate-intensity continuous exercise (Experimental): Moderate-intensity continuous exercise training
  Interventions: Behavioral: moderate-intensity continuous exercise training
- High-Intensity Interval Training (Experimental): High-Intensity Interval Training
  Interventions: Behavioral: high-intensity interval training

INTERVENTIONS:
Behavioral: moderate-intensity continuous exercise training — Participants will complete supervised exercise sessions. Moderate-intensity continuous exercise training will follow cardiovascular rehabilitation guidelines. Participants will attend on-site moderate-intensity continuous exercise training two times weekly for 12 weeks.
  Arms: Moderate-intensity continuous exercise
Behavioral: high-intensity interval training — Participants will complete supervised exercise sessions. Participants will attend on-site high-intensity interval training two times weekly for 12 weeks.
  Arms: High-Intensity Interval Training

SUMMARY:
Atrial fibrillation is the most common heart rhythm disorder. The management of atrial fibrillation is of great importance. Despite the presence of exercise intolerance, weight gain, and an associated decline in overall health and well-being in patients living with atrial fibrillation, recommended standard care does not currently include the prescription of exercise to address these significant health issues. Exercise training is a recognized form of treatment of persons with heart disease. An exercise program such as high-intensity interval training when compared to moderate-intensity continuous exercise training may provide a stronger training stimulus for exercise and clinical outcomes; may be more efficient and motivating; and, may help to improve adherence to exercise training in persistent or permanent atrial fibrillation patients. This has been shown in patients with coronary artery disease and heart failure.

The primary objectives of this prospective study are to examine the impact of high-intensity interval training compared to moderate-intensity continuous exercise training in adults with persistent or permanent atrial fibrillation on exercise capacity and quality of life.

DETAILED DESCRIPTION:
Atrial fibrillation is the most common heart rhythm disorder. Significant disease and death rates are associated with atrial fibrillation because of stroke risk, the complications of medications, poor quality of life and reduced exercise tolerance. Many patients report they have a lower quality of life because of this condition, so finding new ways of helping patients manage and cope with this health problem may help a great number of people. The management of atrial fibrillation is of great importance. Despite the presence of exercise intolerance, weight gain, and an associated decline in overall health and well-being in patients living with atrial fibrillation, recommended standard care does not currently include the prescription of exercise to address these significant health issues. Exercise training is a recognized form of treatment of persons with heart disease. An exercise program such as high-intensity interval training when compared to moderate-intensity continuous exercise training may provide a stronger training stimulus for exercise and clinical outcomes; may be more efficient and motivating; and, may help to improve adherence to exercise training in persistent or permanent atrial fibrillation patients. This has been shown in patients with coronary artery disease and heart failure.

The primary objectives of this prospective study are to examine the impact of high-intensity interval training compared to moderate-intensity continuous exercise training in adults with persistent or permanent atrial fibrillation on exercise capacity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. persistent or permanent atrial fibrillation;
2. rate controlled with a resting ventricular rate of equal to or less than 110 bpm;
3. able to perform a symptom-limited exercise test;
4. at least 40 years of age;
5. patient agrees to sign informed consent.

Exclusion Criteria:

1. currently participating in routine exercise training (more than two times per week);
2. unstable angina;
3. uncontrolled diabetes mellitus;
4. diagnosed severe mitral or aortic stenosis;
5. diagnosed hypertrophic obstructive cardiomyopathy with significant obstruction;
6. unable to provide written, informed consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-11; Primary Completion 2030-01 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life as measured by the Short-Form 36 questionnaire | baseline to 12 weeks
  Change in quality of life from baseline to 12 weeks as measured by the Short Form-36 questionnaire.
Change in exercise capacity as measured by six-minute walk test distance | baseline to 12 weeks
  Change in exercise capacity from baseline to 12 weeks as measured by six-minute walk test distance.

SECONDARY OUTCOMES:
Change in exercise adherence measured by accelerometer | baseline to 12 weeks
  Change in exercise adherence from baseline to 12 weeks as measured by accelerometer.
Change in activity status measured by the Duke Activity Status Index | baseline to 12 weeks
  Change in activity status from baseline to 12 weeks as measured by the Duke Activity Status Index.
Change in symptom burden measured by the Canadian Cardiovascular Society Severity of Atrial Fibrillation scale | baseline to 12 weeks
  Change in symptom burden from baseline to 12 weeks as measured by the Canadian Cardiovascular Society Severity of Atrial Fibrillation scale.
Change in symptom frequency and severity measured using the 7-day symptom diary | baseline to 12 weeks
  Change in symptom frequency and severity from baseline to 12 weeks as measured using the the 7-day symptom diary.
Change in disease specific quality of life will be measured using the University of Toronto Atrial Fibrillation Severity Scale (AFSS) | baseline to 12 weeks
  Change in disease specific quality of life from baseline to 12 weeks will be measured using the University of Toronto Atrial Fibrillation Severity Scale (AFSS).
Change in anxiety and depressive symptoms will be measured using the Hospital Anxiety and Depression Scale (HADS) | baseline to 12 weeks
  Change in anxiety and depressive symptoms from baseline to 12 weeks will be measured using the Hospital Anxiety and Depression Scale (HADS).
Change in sleep apnea risk will be measured by the STOP-BANG Sleep Apnea Questionnaire | baseline to 12 weeks
  Change in risk of sleep apnea from baseline to 12 weeks will be measured by the STOP-BANG Sleep Apnea Questionnaire.
Insomnia severity index will be measured using the Insomnia Severity Index | baseline to 12 weeks
  Insomnia severity index at baseline and 12 weeks will be measured using the Insomnia Severity Index.
Change in self reported sleep patterns will be measured using a 7-day sleep diary | baseline to 12 weeks
  Change in self reported sleep patterns from baseline to 12 weeks will be measured using a 7-day sleep diary.
Change in heart rate control will be measured using 24-hour Holter ECG recordings and ECG recordings at each cardiopulmonary exercise test (CPET) | baseline to 12 weeks
  Change in heart rate control from baseline to 12 weeks will be measured using 24-hour Holter ECG recordings and ECG recordings at each cardiopulmonary exercise test (CPET)
Change in muscular fitness will be measured using standard load tests | baseline to 12 weeks
  Change in muscular fitness from baseline to 12 weeks will be measured using standard load tests.
Change in exercise capacity will be measured using a cardiopulmonary exercise test (CPET) | baseline to 12 weeks
  Change in exercise capacity from baseline to 12 weeks will be measured using a cardiopulmonary exercise test (CPET)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Reed, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Insititue, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Reed JL, Terada T, Vidal-Almela S, Tulloch HE, Mistura M, Birnie DH, Wells GA, Nair GM, Hans H, Way KL, Chirico D, O'Neill CD, Pipe AL. Effect of High-Intensity Interval Training in Patients With Atrial Fibrillation: A Randomized Clinical Trial. JAMA Netw Open. 2022 Oct 3;5(10):e2239380. doi: 10.1001/jamanetworkopen.2022.39380. PMID 36315143